CLINICAL TRIAL: NCT04817878
Title: Cohort Construction for Preterm Infants With Growth Retardation and Its Influencing Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Xiaomei Tong, Director, Head of peadiatrics, Clinical Professor, Peking University Third Hospital
Other Study IDs: bysy2020-423-01
Record Dates: First submitted 2021-03-16; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Problem With Growth of an Infant
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood routine， Convenience routine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Late preterm infant group: Gestational age 33 weeks-36 weeks
  Interventions: Combination Product: Developmental assessment
- Very premature infant group: Gestational age 28 weeks-32 weeks
  Interventions: Combination Product: Developmental assessment
- Super preterm infant group: Gestational age less than 28 weeks
  Interventions: Combination Product: Developmental assessment

INTERVENTIONS:
Combination Product: Developmental assessment — Physical development assessment (head circumference, length, weight), Neurodevelopment assessment at 36 to 40 weeks of correction (GMS assessment, NBNA assessment), neurodevelopment assessment at 18 months, 24 months, and 36 months (ASQ scale, Language assessment, Wei-style scale), audiovisual screening, etc.

SUMMARY:
In this cohort, prospective clinical cohort study was used to establish a follow-up cohort of preterm infants with different gestational ages. The regular monitoring indexes of physical development and neuropsychological development of preterm infants from birth to 3 years after birth were collected. The influencing factors of preterm infants' development at different stages were recorded, and the high-risk factors leading to different stages of preterm infants' growth retardation were analyzed.

DETAILED DESCRIPTION:
Preterm infants are at high risk of stunting due to premature birth, insufficient intrauterine nutrient reserves, burden of various diseases after birth, and persistent nutrient liabilities. The growth retardation of premature infants at different developmental stages has an important impact on both short-term survival and long-term health. The growth and development data of premature infants during hospitalization and after discharge are very limited in foreign countries. Domestic researches on growth retardation of preterm infants only involve retrospective cross-sectional studies during hospitalization, and lack of prospective follow-up study data on growth and development data of premature infants during hospitalization and after discharge.

In this cohort, prospective clinical cohort study was used to establish a follow-up cohort of preterm infants with different gestational ages. The regular monitoring indexes of physical development and neuropsychological development of preterm infants from birth to 3 years after birth were collected. The influencing factors of preterm infants' development at different stages were recorded, and the high-risk factors leading to different stages of preterm infants' growth retardation were analyzed. In order to provide a strong scientific basis for the development evaluation and intervention of premature infants in China, a systematic and scientific clinical cohort study method was explored to improve the overall medical quality and medical level of the Department and further promote the development of the discipline.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants born less than 37 weeks during the study period

Exclusion Criteria:

* Congenital malformations or genetic diseases Various surgical treatments during the newborn period Interrupted treatment or discharged automatically

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants born during the study period
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of extrauterine growth retardation of preterm infants at 36-40 weeks of gestational age correction | correct gestational age 36~40 weeks
  According to Fenton 2003 growth curve of premature infants, the weight, length, and head circumference of preterm infants with corrected gestational age of 36-40 weeks were evaluated, If the weight, length and head circumference are lower than the 10th percentile of the corresponding gestational age, the child is diagnosed as EUGR（extrauterine growth retardation）
Assessment of neurodevelopmental retardation of preterm infants at 36-40 weeks of gestational age correction | correct gestational age 36~40 weeks
  IF the NBNA score of preterm infants at 36-40 weeks of correction is lower than 36, and the abnormal GMs is evaluated, the child is diagnosed as neurodevelopmental retardation.
Assessment of low weight of preterm infants at 2 to 3 years of age | 2~3 years old
  Compared with the same age and gender reference population standard, children's weight below the median minus 2 standard deviations (i.e. less than the 3rd percentile) is diagnosed as low weight
Assessment of growth retardation of preterm infants at 2 to 3 years of age | 2~3 years old
  Compared with the same age and gender reference population standard, children's height below the median minus 2 standard deviations (i.e. less than the 3rd percentile) is diagnosed as growth retardation
Assessment of small head circumference of preterm infants at 2 to 3 years of age | 2~3 years old
  Compared with the same age and gender reference population standard, the children's occipitofrontal circumference (OFC) less than 2 standard deviations (SD) of the mean OFC (i.e. less than the 3rd percentile) is diagnosed as small head circumference
Assessment of neurodevelopmental retardation of preterm infants at 2 to 3 years of age | 2~3 years old
  IF the Wechsler intelligence scales score is lower than 70, the child is diagnosed as neurodevelopmental retardation.

CONTACTS AND LOCATIONS:
Overall Officials: xiaomei tong, Ph.D., Principal Investigator — Peking University Third Hospital; yanmei chang, Ph.D., Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China